CLINICAL TRIAL: NCT04995276
Title: PostmenopausAL heaLth And DIseAse (PALLADIA) Study: Prospective Study of the Incidence and Risk Factors of Chronic Diseases Associated With Menopause
Brief Title: PostmenopausAL heaLth And DIseAse (PALLADIA) Study
Acronym: PALLADIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Irene Lambrinoudaki, Professor of Endocrinology, National and Kapodistrian University of Athens
Other Study IDs: 8259
Record Dates: First submitted 2021-07-23; First posted 2021-08-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Menopause
Keywords: menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

SUMMARY:
This is a prospective study of the incidence and risk factors of chronic diseases that are associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women

Exclusion Criteria:

Men Women of reproductive age

Ages: 15 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postmenopausal women
Study Population: The study will include 4.000 postmenopausal women
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | up to 2025
Coronary heart disease | up to 2025
Stroke | up to 2025

SECONDARY OUTCOMES:
Diabetes mellitus | up to 2025
Osteoporotic fractures | up to 2025
Breast cancer | up to 2025
Any cancer | up to 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Menopause Clinic, Aretaieio Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No